CLINICAL TRIAL: NCT06683287
Title: Effects of Low-Level Red Light and Distant-Image Screen for Myopia Control in Children: a Randomized Controlled Trial
Brief Title: Effects of Low-Level Red Light and Distant-Image Screen for Myopia Control in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, cao kai, Dr, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BeijingTH2024qiao
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Myopia
Keywords: myopia; red-light; distant-image screen
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- red-light (Experimental): Children in this group received a red-light apparatus (LS-03B; Yishiliang Inc), which has been deemed safe by the State Administration for Market Regulation of China. They were directed to utilize this apparatus twice a day for 3-minute sessions, ensuring a gap of over 4 hours between each use.
  Interventions: Device: red light
- distant-image screen group (Experimental): participants were given a distant-image screen ( RIO-Max2.0; Ruishi Inc), and were asked to use this device for ≥1 hour/day
  Interventions: Device: distant image screen
- red-light plus distant image screen (Experimental): For this group, participants were given a red-light device (LS-03B; Yishiliang Inc) and a distance image screen device ( RIO-Max2.0; Ruishi Inc), and were asked to use red-light twice a day for 3-minute sessions, ensuring a gap of over 4 hours between each use, and use distant image screen for ≥1 hour/day
  Interventions: Device: red light and distant image screen
- control (No Intervention): No intervention

INTERVENTIONS:
Device: red light and distant image screen — red light plus distant image screen, children use these two devices at the same time
  Arms: red-light plus distant image screen
Device: red light — children use red light for 3 minutes each time, twice a day
  Arms: red-light
Device: distant image screen — Children in this group were asked to use this device for ≥1 hour/day
  Arms: distant-image screen group

SUMMARY:
This study aims to assess the efficacy and safety of daily exposure to 650-nm low-level red light (RL) and distant-image therapy (DIT) for myopia treatment.

DETAILED DESCRIPTION:
This was a randomized clinical trial. Children aged 8 to 10 years with a spherical equivalent error (SER) ranging from -1 to -1.5 diopters (D) were enrolled, and were randomly allocated to the following treatment group: RL, DIT, RL plus DIT, and control in a 1:1:1:1 ratio. The primary outcomes were one-year change in SER and axial length.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age between 8 and 10 years old. 2. The spherical equivalent error after pupil dilation was between -1.0 D and -1.5D.

  3. Corneal astigmatism ≤ 1.25D. 4. Interocular refraction discrepancy ≤ 1.5D. 5. Near-distance exophoria < 10 prism diopters (△) and far-distance exophoria < 6 prism diopters (△).

  6. Willingness to participate in the study and signed informed consent.

Exclusion Criteria:

* 1. Intraocular pressure was below 10 mmHg or higher than 22 mm Hg. 2. Presence of amblyopia, or ocular pathological conditions such as retinal, lens, or corneal disorders.

  3. Children currently using atropine or orthokeratology for myopia control. 4. Patients with systemic and immune disorders such as albinism, psoriasis, nephrotic syndrome, systemic lupus erythematosus, diabetes, etc.

  5. Individuals with conditions like Tourette's syndrome or epilepsy.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Changes in axial length | one year
  Axial length was measured using an optical biometer (Colombo IOL, Moptim)
Changes in spherical equivalent error | one year
  Spherical equivalent error was calculated from the dioptric powers of the sphere and half of the cylinder.The children's pupils were dilated using tropicamide eyedrops, then SER was subsequently measured using an auto refractor (ARK-510A, Nidek Co Ltd)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, China, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang K, Wang Y, Li X, Liu S, Shi H, Qiao L. One-year changes in axial length and refraction in children using low-level red light and distant-image screen for myopia control: a randomized controlled trial. Front Med (Lausanne). 2025 Mar 25;12:1542620. doi: 10.3389/fmed.2025.1542620. eCollection 2025. PMID 40201319